CLINICAL TRIAL: NCT02013414
Title: Molecular Image-directed, 3D Ultrasound-guided Biopsy of the Prostate
Brief Title: Fusion Targeted Biopsy of the Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Baowei Fei, PhD, EngD, Associate Professor and Georgia Cancer Coalition Dinstinguished Cancer Scholar, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00045065; R01CA156775 (NIH); R21CA176684 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2013-12-17 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 3D ultrasound-guided biopsy (Experimental): Participants will have a 3D ultrasound-guided biopsy of the prostate rather than the standard of care 2D ultrasound-guided biopsy.
  Interventions: Device: 3D ultrasound-guided biopsy

INTERVENTIONS:
Device: 3D ultrasound-guided biopsy — Patients will have a PET/CT prior to the biopsy. The CT images will be combined with the PET images for improved localization of suspicious tumors. During the biopsy, the 3-D ultrasound images will be acquired immediately before the biopsy while the patient is on the table. The ultrasound images together with the PET images will be used to guide the targeted biopsy of the prostate.

SUMMARY:
The objective of the proposed study is to evaluate a new, molecular image directed, three-dimensional (3D) ultrasound guided biopsy system in human patients. The current biopsy uses ultrasound imaging as guidance. However, the procedure uses two-dimensional (2D) ultrasound images and has sampling errors thus some cancers can be missed from the standard 2D image-guided biopsy. In this study, an FDA-approved ultrasound device will be used to obtain three-dimensional (3D) images of the prostate from a commercially available ultrasound scanner. The clinician can use the 3D images to guide biopsy, record the core location of the biopsy sites, and perform re-biopsy to the same sites in a patient follow-up examination. This system can also use images from magnetic resonance imaging (MRI) or positron emission tomography (PET) and then fuse PET or MR images with 3D ultrasound images to guide the needle to a suspicious tumor target as seen on MRI or PET. We think that this fusion targeted biopsy technology will help to improve the accuracy of the current systematic biopsy approach for prostate cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older
* Abnormal uptake in prostate necessitating a biopsy
* Able to provide informed consent

Exclusion Criteria:

* Age less than 18
* Cannot provide informed consent
* Less than 2 months since any prior prostate biopsy (to decrease false positive uptake from inflammation)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baowei Fei, PhD, EngD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Targeted Biopsy and Template Biopsy: Study participants with abnormal FACBC PET-CT scans received a fluciclovine PET ultrasound fusion targeted biopsy and a template (standard of care) biopsy to test the feasibility of targeted biopsies for detecting recurrent prostate cancer.
Period: Overall Study
Arm/Group | Targeted Biopsy and Template Biopsy
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Targeted Biopsy and Template Biopsy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.08 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Cancer Detection by Targeted and Standard Biopsy Approaches
Description: The feasibility of detecting cancer detection with the targeted prostate biopsy was assessed. This study sought only to determine if the targeted biopsy approach was able to detect recurrent prostate cancer and values for the number of samples testing positive for cancer per each biopsy approach are not available. This feasibility study preceded a clinical trial (NCT02744534) assessing the accuracy of prostate cancer detection with targeted biopsies compared to the standard biopsy.
Time Frame: Up to 2 years
Population: Only whether or not the targeted biopsy could detect cancer was examined and the number of positive biopsy cores per each biopsy approach were not determined.
Groups:
- Targeted Biopsy: Fluciclovine defined targets were biopsied using the 3-D visualization and navigation platform to guide the biopsy needle and record its path
- Standard Biopsy: The standard transrectal ultrasound guided biopsy collects 2 cores per region (when possible) from 6 standard regions of the prostate.
Arm/Group | Targeted Biopsy | Standard Biopsy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: As adverse events related to the radiotracer injection were not expected, adverse events were not collected for this feasibility study.
Description: Adverse events were not collected thus the number of participants at risk is zero.
Arm/Group | Targeted Biopsy | Standard Biopsy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-07-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT02013414/Prot_000.pdf